CLINICAL TRIAL: NCT02271269
Title: A Randomized Controlled Trial to Increase Glaucoma Medication Adherence Using Value Pricing
Brief Title: Study on Incentives for Glaucoma Medications Adherence
Acronym: SIGMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Marcel Bilger, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSRNIG12nov007
Record Dates: First submitted 2014-10-19; First posted 2014-10-22 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Glaucoma
Keywords: glaucoma; medication adherence; financial incentives; behavioral economics
MeSH Terms: conditions — Glaucoma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (UC) (No Intervention): Patients receiving Usual Care for Glaucoma comprising:
  * Education on effective glaucoma treatment
  * Routine check-ups with an ophthalmologist and prescription of glaucoma eye drops
  * Glaucoma counselling [Can be recommended by ophthalmologist for non-adherent patients] covering:
    * Glaucoma risk factors and symptoms
    * Management and treatment
    * Medications and optimal dosage windows
    * Risks of medication non-adherence
    * Formulation of a dosing schedule that compliments each patient's lifestyle
- Value Pricing (VP) (Experimental): Patient receiving Usual Care for Glaucoma and given the opportunity to receive Value Pricing Subsidies.
  Interventions: Behavioral: Value Pricing Subsidies

INTERVENTIONS:
Behavioral: Value Pricing Subsidies — * Usual care for glaucoma
  * Subsidies granted to adherent patients for their glaucoma medications and physician visits, lowering the costs of treatment and providing a financial incentive for patients to take their medicines as prescribed.
  * Subsidy (25 / 50%) granted based on meeting dose-rate adherence percentage targets (75 / 90%) at the month 3 and 6 assessment points.
  Arms: Value Pricing (VP)

SUMMARY:
Glaucoma topical eye medications, when adhered to, are effective at controlling disease progression. Yet evidence shows that many glaucoma patients have incomplete adherence to medications, with disease progression resulting in significant costs to the patient and health system. Through the approach of value pricing, a link can be made between non-adherence and its resulting costs by granting subsidies to adherent patients for their medications and physician visits. This 6-month randomized controlled trial among 100 glaucoma patients from the Singapore National Eye Centre aims to test the extent to which value pricing can improve medication adherence.

DETAILED DESCRIPTION:
By reducing intraocular pressure, glaucoma topical eye medications are effective at controlling disease progression for the majority of patients. Yet evidence shows that many glaucoma patients have incomplete adherence to medications, resulting in significant personal costs in terms of disease progression and visual field loss. The cost to the health system from poor adherence is also substantial as glaucoma surgery is more costly than treatment with topical medication. Behavioural economics theory suggests that adherence rates can be improved by providing a clearer link between non-adherence and the resulting costs thereof. In the proposed study, this link is made by granting subsidies to adherent patients for their medications and physician visits, whereas those who are not sufficiently adherent would not receive the subsidy and thus pay a higher rate for their treatment.

These subsidies provide a financial incentive for patients to take their medicines as prescribed, and because prescription refills and visits occur regularly, also provide a tangible and near-term cost resulting from non-adherence. The investigators refer to this approach as value pricing as subsidies are allocated to medications that have not only been shown to be clinically effective but that are also effectively used by the patient. In efforts to increase adherence among glaucoma patients in Singapore, the investigators propose to conduct a 6-month proof-of-concept randomized controlled trial among 100 participants from the Singapore National Eye Centre (SNEC) to test the extent to which value pricing can improve medication adherence. As Singapore's population continues to age and a larger share of the population requires daily medications to treat chronic diseases, such innovative solutions are needed to ensure not only that patients take their medications as prescribed and receive the full benefit of their treatment but also that Government subsidies are allocated effectively so that to ensure the sustainability of the health system.

Specific Aim and hypothesis tested:

Aim: Test whether adding Value Pricing (VP) to Usual Care (UC) can improve medication adherence over a 6-month period.

Hypothesis: VP patients will show greater adherence rates at 6 months compared to those receiving only UC.

ELIGIBILITY:
Inclusion Criteria:

* Singaporean citizens or permanent residents
* Conversant in English or Mandarin
* Taking at least one glaucoma eye drop medication
* Shown to be non-adherent based on a value of 6 or less on the Modified Medication Adherence Scale (MMAS)

Exclusion Criteria:

* Significant comorbid conditions preventing application of medications without assistance
* Stage 4 (advanced) or Stage 5 (end stage) glaucoma according to the Glaucoma Staging System

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Monthly dose-rate adherence percentage | Month 6
  The proportion of days across a month where a patient took all medication(s) within the appropriate dosing windows (morning, afternoon, evening) for the day.

SECONDARY OUTCOMES:
Dose-rate adherence percentage | Months 1 - 6
  The proportion of days across the study period where a patient took all medication(s) within the appropriate dosing windows (morning, afternoon, evening) for the day.
Proportion meeting 90% dose-rate adherence percentage | Months 3 & 6
  The proportion of participants at each time point who met the 90% dose-rate adherence percentage cut-off for each monitoring period.
Proportion meeting 75% dose-rate adherence percentage | Months 3 & 6
  The percentage of participants at each time point who met the 75% dose-rate adherence percentage cut-off for each monitoring period.
Intraocular Pressure | Baseline & Month 6
  Intraocular Pressure measured using established protocols at SNEC.
EQ-5D-5L | Baseline & Month 6
  Scale to assess health related quality of life.
Glaucoma Quality of Life (GQL-15) | Baseline & Month 6
  Scale to measure quality of life, pertaining specifically to aspects of QoL that can be affected by the glaucoma condition.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Bilger, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Singapore National Eye Center, Singapore, Singapore

REFERENCES:
- [Background] Elliott RA, Shinogle JA, Peele P, Bhosle M, Hughes DA. Understanding medication compliance and persistence from an economics perspective. Value Health. 2008 Jul-Aug;11(4):600-10. doi: 10.1111/j.1524-4733.2007.00304.x. Epub 2008 Jan 8. PMID 18194403
- [Background] Chapman GB, Brewer NT, Coups EJ, Brownlee S, Leventhal H, Leventhal EA. Value for the future and preventive health behavior. J Exp Psychol Appl. 2001 Sep;7(3):235-50. PMID 11676102
- [Background] van Dulmen S, Sluijs E, van Dijk L, de Ridder D, Heerdink R, Bensing J. Patient adherence to medical treatment: a review of reviews. BMC Health Serv Res. 2007 Apr 17;7:55. doi: 10.1186/1472-6963-7-55. PMID 17439645
- [Background] Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000011. doi: 10.1002/14651858.CD000011.pub3. PMID 18425859
- [Background] Giuffrida A, Torgerson DJ. Should we pay the patient? Review of financial incentives to enhance patient compliance. BMJ. 1997 Sep 20;315(7110):703-7. doi: 10.1136/bmj.315.7110.703. PMID 9314754
- [Background] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Mills RP, Budenz DL, Lee PP, Noecker RJ, Walt JG, Siegartel LR, Evans SJ, Doyle JJ. Categorizing the stage of glaucoma from pre-diagnosis to end-stage disease. Am J Ophthalmol. 2006 Jan;141(1):24-30. doi: 10.1016/j.ajo.2005.07.044. PMID 16386972
- [Background] Horne R, Weinman J. Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness. J Psychosom Res. 1999 Dec;47(6):555-67. doi: 10.1016/s0022-3999(99)00057-4. PMID 10661603
- [Background] Tsai JC, McClure CA, Ramos SE, Schlundt DG, Pichert JW. Compliance barriers in glaucoma: a systematic classification. J Glaucoma. 2003 Oct;12(5):393-8. doi: 10.1097/00061198-200310000-00001. PMID 14520147
- [Derived] Bilger M, Wong TT, Lee JY, Howard KL, Bundoc FG, Lamoureux EL, Finkelstein EA. Using Adherence-Contingent Rebates on Chronic Disease Treatment Costs to Promote Medication Adherence: Results from a Randomized Controlled Trial. Appl Health Econ Health Policy. 2019 Dec;17(6):841-855. doi: 10.1007/s40258-019-00497-0. PMID 31317511
- [Derived] Bilger M, Wong TT, Howard KL, Lee JY, Toh AN, John G, Lamoureux EL, Finkelstein EA. Study on Incentives for Glaucoma Medication Adherence (SIGMA): study protocol for a randomized controlled trial to increase glaucoma medication adherence using value pricing. Trials. 2016 Jul 15;17(1):316. doi: 10.1186/s13063-016-1459-1. PMID 27422389